CLINICAL TRIAL: NCT03974919
Title: Preoperative Pulmonary Systolic Pressure and Outcome After Non-Cardiac Surgery:Threshold Analysis
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Yan Zhou, MD, Principal Investigator, Peking University First Hospital
Other Study IDs: MAEPSP
Record Dates: First submitted 2019-06-03; First posted 2019-06-05 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Hypertension, major cardiovascular event, non-cardiac surgery,threshold
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: NO intervention required — NO intervention required

SUMMARY:
The linear or nonlinear relationship of pulmonary systolic pressure and cardiovascular and kidney outcome after non-cardiac surgery is unknown. This study is to explore the relationship of the two and try to identify the possible threshold of pulmonary systolic pressure for major cardio-vascular events after non-cardiac surgery.

DETAILED DESCRIPTION:
The linear or nonlinear relationship of pulmonary systolic pressure and cardiovascular and kidney outcome after non-cardiac surgery is unknown. This study is to explore the relationship of the two and try to identify the possible threshold of pulmonary systolic pressure for major cardio-vascular events after non-cardiac surgery.

Patients with preoperative cardio-echogram under going non-cardiac surgery were collected. The postoperative major cardiovascular, cerebral and kidney events were also identified and collected. Other data including peri-operative information and surgeries and anesthesia data were gathered.

Logistic regression models were built and selected. Independent risk factors relative to postoperative major cardiovascular and cerebral events were screened and identified. Odds ratio, relative risk and relative risk ratio of varies dichomitus cut points were calculated, trend breakpoint were identified, propensity score analysis were also done for causal inference.

ELIGIBILITY:
Inclusion Criteria:

non-cardiac surgery patients with preoperative echocardiography records

Exclusion Criteria:

electronic records missing or peri-operative data missing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: non-cardiac surgery adult patients with preoperative echocardiography
Sampling Method: Non-Probability Sample
Enrollment: 19000 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-11 (Actual)

PRIMARY OUTCOMES:
major adverse events | 30 days postoperatively in hospital
  cardiac infarction, heart failure, cardiac death, stroke, acute kidney injury

CONTACTS AND LOCATIONS:
Locations (1):
- First hospital Peking University, Beijing, Beijing Municipality, China